CLINICAL TRIAL: NCT04314661
Title: Innovative Osteoarthritis Therapy Using Combination of Mesenchymal Stem Cell (MSC) and Conditioned Medium (CM): A Comparative Study on Arthroscopy and Non-Arthroscopy
Brief Title: Mesenchymal Stem Cell Therapy (MSCs) and Conditioned Medium Therapy for Osteoartrithis
Acronym: OA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/OA/02/2022
Record Dates: First submitted 2020-02-19; First posted 2020-03-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Allogeneic Mesenchymal Stem Cells; Umbilical Cord; Conditioned Medium
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroscopy; Secretome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arthroscopy + Booster (Experimental): After arthroscopy intervention, patient will be given 10 million UC-MSCs and 2 cc Secretome twice with 2 weeks interval via intra-articular injection.
  Interventions: Biological: Arthroscopy with Mesenchymal Stem Cells + Secretome + Secretome
- Arthroscopy + Pre-Conditioning (Experimental): After arthroscopy intervention, patient will be given 2 cc Secretome, 10 million UC-MSCs, and 2 cc Secretome with 2 weeks interval via intra-articular injection.
  Interventions: Biological: Arthroscopy with Secretome + Mesenchymal Stem Cells + Secretome
- Non Arthroscopy + Booster (Experimental): Without arthroscopy intervention, patient will be given 10 million UC-MSCs and 2 cc Secretome twice with 2 weeks interval via intra-articular injection.
  Interventions: Biological: Non Arthroscopy with Mesenchymal Stem Cells + Secretome + Secretome
- Non Arthroscopy + Pre-Conditioning (Experimental): Without arthroscopy intervention, patient will be given 2 cc Secretome, 10 million UC-MSCs, and 2 cc Secretome with 2 weeks interval via intra-articular injection.
  Interventions: Biological: Non Arthroscopy with Secretome + Mesenchymal Stem Cells + Secretome

INTERVENTIONS:
Biological: Arthroscopy with Mesenchymal Stem Cells + Secretome + Secretome — After Arthroscopy intervention, patient recieve 10 million Allogeneic Umbilical Cord Mesenchymal Stem Cells in 2 cc NaCl, two weeks afterward, patient receive 2 cc Secretome, and four weeks later, patient receive another 2 cc Secretome. All intervention will be done via Intra-articular.
  Arms: Arthroscopy + Booster
Biological: Arthroscopy with Secretome + Mesenchymal Stem Cells + Secretome — After Arthroscopy intervention, patient recieve 2 cc Secretome, two weeks afterward patient receive 10 million Allogeneic Umbilical Cord Mesenchymal Stem Cells in 2 cc NaCl, and four weeks later, patient receive another 2 cc Secretome. All intervention will be done via Intra-articular.
  Arms: Arthroscopy + Pre-Conditioning
Biological: Non Arthroscopy with Mesenchymal Stem Cells + Secretome + Secretome — Without Arthroscopy intervention, patient recieve 10 million Allogeneic Umbilical Cord Mesenchymal Stem Cells in 2 cc NaCl, two weeks afterward, patient receive 2 cc Secretome, and four weeks later, patient receive another 2 cc Secretome. All intervention will be done via Intra-articular.
  Other Names: Secretome
  Arms: Non Arthroscopy + Booster
Biological: Non Arthroscopy with Secretome + Mesenchymal Stem Cells + Secretome — Without Arthroscopy intervention, patient recieve 2 cc Secretome, two weeks afterward patient receive 10 million Allogeneic Umbilical Cord Mesenchymal Stem Cells in 2 cc NaCl, and four weeks later, patient receive another 2 cc Secretome. All intervention will be done via Intra-articular.
  Arms: Non Arthroscopy + Pre-Conditioning

SUMMARY:
This study aims to compare the efficacy of Umbilical Cord Mesenchymal Stem Cell and secretome between arthroscopy and without arthroscopy intervention in OA patients. This study has 4 arms namely Arthroscopy + Booster, Arthroscopy + Pre-conditioning, Non-Arthroscopy + Booster, Non-Arthroscopy + Pre-conditioning.

DETAILED DESCRIPTION:
The study subjects each group amounted to 5 patients suffering from osteoarthritis. Patients are evaluated before, and 1,3,6 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 55-70 years
* Suffering from grade 2-3 OA was identified by two observers who differed accordingly Kellgren-Lawrence research scale
* Absence of local or general infections
* Haematological and biochemical analysis without significant changes being made cause contraindications
* Patients can understand the nature of the study
* Written informed consent is given to patients

Exclusion Criteria:

* Patients are not willing to obey the study protocol
* There are signs of infection or positive serology for HIV, hepatitis and syphilis
* There is a history of cancer both in the family and yourself and the value of the examination tumour marker exceeds normal limits
* There is a congenital disease that causes significant deformity of the knee can interfere with cell applications and interpret results
* Articular injection of the knee by any drug during the previous 3 months
* Participate in any clinical trial or treatment 30 days before the study
* Other conditions may, according to medical criteria, not support participation in this research
* Patients are subordinates or low ranking members

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-07-08 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 1 month after injection
  To asses pain score, score 1(good)-10(worst)
Visual Analog Scale (VAS) | 3 month after injection
  To asses pain score, score 1(good)-10(worst)
Visual Analog Scale (VAS) | 6 month after injection
  To asses pain score, score 1(good)-10(worst)
Western Ontario and McMaster Universities Osteoarthritis Index | 1 month after injection
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints.
Western Ontario and McMaster Universities Osteoarthritis Index | 3 month after injection
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints.
Western Ontario and McMaster Universities Osteoarthritis Index | 6 month after injection
  To evaluate the condition of patients with osteoarthritis, including pain, stiffness, and physical functioning of the joints.

SECONDARY OUTCOMES:
Laboratory Asessment | 2 weeks after injection
  COMP, MMP-13, IL-6
Laboratory Asessment | 1 month after injection
  COMP, MMP-13, IL-6
Laboratory Asessment | 3 months after injection
  COMP, MMP-13, IL-6
Magnetic Resonance Imaging (MRI) T2 mapping | 6 month after injection
  MRI T2 mapping is used for cartilage evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Gatot Soebroto Hospital, Jakarta Pusat, DKI Jakarta, Indonesia